CLINICAL TRIAL: NCT05064735
Title: Effect of Subcutaneous Semaglutide 2.4 mg Once-weekly Compared to Placebo in Subjects With Obesity and Knee Osteoarthritis
Brief Title: Research Study Looking at How Well Semaglutide Works in People Suffering From Obesity and Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NN9536-4578; U1111-1246-5824 (Other: WHO); 2020-000204-11 (EudraCT Number)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- semaglutide 2.4 mg (Experimental): Participants will receive semaglutide subcutaneous (s.c) 2.4 mg once-weekly as adjunct to a reduced-calorie diet and increased physical activity
  Interventions: Drug: semaglutide 2.4 mg
- semaglutide 2.4 mg (placebo) (Placebo Comparator): Participants will receive semaglutide subcutaneous (s.c) placebo once-weekly as adjunct to a reduced-calorie diet and increased physical activity
  Interventions: Drug: semaglutide 2.4 mg (placebo)

INTERVENTIONS:
Drug: semaglutide 2.4 mg — semaglutide subcutaneous (s.c.) 2.4 mg once-weekly or semaglutide placebo once-weekly as adjunct to a reduced-calorie diet and increased physical activity
  Arms: semaglutide 2.4 mg
Drug: semaglutide 2.4 mg (placebo) — semaglutide subcutanous (s.c.) 2.4 mg once-weekly or semaglutide placebo once-weekly as adjunct to a reduced-calorie diet and increased physical activity
  Arms: semaglutide 2.4 mg (placebo)

SUMMARY:
This study will look at participants body weight from the start to the end of the study. It will also look at how much pain participants have in participants knee from the start to the end of the study and how this affects participants daily life. This is to compare the effect on body weight and pain in the knee in people taking semaglutide with people taking "dummy" medicine. Participants will either get semaglutide or "dummy" medicine. Which treatment participants get is decided by chance.

Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. During the study, participants will have talks with study staff about how to eat healthy food and how to be more physically active. The study will last for about 1 ½ years. Participants will have 14 clinic visits with the study staff. At the first clinic visit participants will have a blood sample taken. Participants will have an X-ray of participants knee taken at the first visit. If participants have had an X-ray recently, this may not be needed.

At 6 of the clinic visits participants cannot take pain medications for 3 days before the visit. Participants cannot take part if participants have had a joint replacement surgery in participants knee. Participants cannot take part if participants have or have had diabetes. Women: Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent
* Body Mass Index (BMI) equal to or greater than 30.0 kg/m^2
* Clinical diagnosis of knee OA (American College of Rheumatology (ACR) criteria) with moderate radiographic changes (Kellgren-Lawrence (KL) grades 2 or 3 as per central reading) in target knee. Target knee joint is defined as most symptomatic knee at screening. If pain in knees are equal target knee joint will be in the most dominant leg.
* Pain due to knee OA

Exclusion Criteria:

* Joint replacement in target knee
* Arthroscopy or injections into target knee within last 3 months prior to enrolment
* Any other joint disease in the target knee

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept. 2834), Study Director — Novo Nordisk A/S
Locations (122):
- United States (61):
  - Baptist Health System, Montgomery, Alabama
  - Ortho Arizona, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Stuart L. Silverman MD - A Medical Corporation, Beverly Hills, California
  - Valley Research, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research of Hollywood_Hollywood, Hollywood, Florida
  - Westside Center For Clinical Research, Jacksonville, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Well Pharma Medical Research Corp, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - East West Medical Research Institute_Honolulu, Honolulu, Hawaii
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Clinical Invest Special_Gurnee, Wauconda, Illinois
  - MediSphere Medical RC, Evansville, Indiana
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - KU MedWest, Shawnee Mission, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Maryland Veterans Administration Health Care System, Baltimore, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Arcturus Healthcare, PLC., Troy, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - The Center For Pharmaceutical Research PC, Kansas City, Missouri
  - Sundance Clinical Research LLC, St Louis, Missouri
  - NYU Langone Medical Cent-Joan H Tisch Cnt for Women's Health, New York, New York
  - Hospital For Special Surgery, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - DaVita Clinical Research - New York, The Bronx, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - University of North Carolina- Chapel Hill Adults, Chapel Hill, North Carolina
  - Medication Mgmnt, LLC_Grnsboro, Greensboro, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Raleigh Medical Group, Raleigh, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Velocity Clin Res_Cincinnati, Cincinnati, Ohio
  - Louis Stokes Clvlnd VA Med Ctr, Cleveland, Ohio
  - Cleveland Clinic_Cleveland, Cleveland, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Altoona Osteoporosis Center, Duncansville, Pennsylvania
  - The University of Penn Center, Philadelphia, Pennsylvania
  - Parkside Family Medicine, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Accellacare US Inc._SC, Mt. Pleasant, South Carolina
  - Coastal Carolina Res Ctr., North Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Tennova HC Turkey Creek MC, Knoxville, Tennessee
  - PrimeCare Medical Group, Houston, Texas
  - Southwest Houston Research Ltd, Houston, Texas
  - DM Clin Rsrch/Fam Diag Clinic, Tomball, Texas
  - Health Res of Hampton Roads, Newport News, Virginia
  - National Clin Res Inc., Richmond, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Canada (16):
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - C-endo Diab & Endo Clinic, Edmonton, Alberta
  - Ocean West Research Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Manna Research Inc. (Burlington N), Burlington, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Dr Anil K Gupta Med Prof Corp, Toronto, Ontario
  - Manna Research Inc._Toronto, Toronto, Ontario
  - Centre Medical Acadie, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
  - Ctr Méd. et pro d l'Ost d port, Saint-Marc-des-Carrieres, Quebec
  - Institut universitaire de cardiologie, Québec
  - Master Centre for Canada, Toronto
- Colombia (4):
  - Centro de investigación médico asistencial S.A.S, Barranquilla
  - BLUECARE SALUD S.A.S. Sede Centro Médico Integral, Bogotá
  - CentrodeInvestigaciónenReumatologíayEspecialidadesMédicas, Bogotá
  - Preventive Care S.A.S, Chía
- Denmark (2):
  - Klinik for Led og bindevævssygdomme, Aarhus N
  - Frederiksberg Hospital - Parker Institutet (Artrose), Frederiksberg
- France (9):
  - Centre Hospitalier de Clermont-Ferrand-Hopital Gabriel Montpied, Clermont-Ferrand
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-2, Le Creusot
  - Aphp-Hopital La Pitie Salpetriere-3, Paris
  - CHU Pitié-Salpétrière, Paris
  - Ap-Hp-Hopital Europeen Georges Pompidou, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hospices Civils de Lyon-Hopital Lyon Sud-1, Pierre-Bénite
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-2, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Norway (3):
  - Akershus Universitetssykehus, Nordbyhagen
  - Oslo us HF, Aker sykehus, Oslo
  - Senter for sykelig overvekt i Helse Sør-Øst, Tønsberg
- Russia (10):
  - PIH "Clin Hosp "RZD-Medicina" former Kazan OJSC Rus Railways, Kazan'
  - LLC Medical center "Maksimum Zdorovia", Kemerovo
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - Setchenov First Moscow State Medical University, Moscow
  - Federal Bureau for Medical and Social Expertise, Moscow
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - SIH "Saratov Regional Clinical Hospital for War Veterans", Saratov
  - Siberian State Medical University, Tomsk
  - Voronezh Regional Clinical Consultive-diagnostic Centre, Voronezh
  - SBCI HC Yaroslavl region "Central City Hospital", Yaroslavl
- Saudi Arabia (4):
  - King Abdulaziz Hospital-Al Ahsa-National Guard, Al Ahsa
  - King Khaled University Hospital,King Saud Univ. Med. City, Riyadh
  - King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh
  - King Fahad Medical City, Riyadh
- South Africa (6):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Dr Wilhase's rooms, Boksburg, Gauteng
  - Chris Hani Baragwanath Hospital, Johannesburg, Gauteng
  - Botho ke Bontle Health Services, Pretoria, Gauteng
  - Dr J Reddy, Durban, KwaZulu-Natal
  - Lenmed Shifa Private Hospital, Durban, KwaZulu-Natal
- Spain (3):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinico San Carlos, Madrid
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
- Sweden (4):
  - Forskningsmottagning Internmedicin (tidigare KFE), Malmo
  - Medicinkliniken Överviktsenheten USÖ, Örebro
  - S:t Göran Sjukhus, Stockholm
  - Department of Metabolism and Endocrinology, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Bliddal H, Bays H, Czernichow S, Udden Hemmingsson J, Hjelmesaeth J, Hoffmann Morville T, Koroleva A, Skov Neergaard J, Velez Sanchez P, Wharton S, Wizert A, Kristensen LE; STEP 9 Study Group. Once-Weekly Semaglutide in Persons with Obesity and Knee Osteoarthritis. N Engl J Med. 2024 Oct 31;391(17):1573-1583. doi: 10.1056/NEJMoa2403664. PMID 39476339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 61 sites in 11 countries as follows (number of sites that screened participants/ number of sites that randomised participants): Canada (5/ 5); Colombia (3/ 3); Denmark (2/ 2); France (5/ 5); Norway (3/ 3); Russia (10/ 10); Saudi Arabia (4/ 4); South Africa (5/ 5); Spain (3/ 3); Sweden (4/ 4) and United States (17/ 17).
Pre-assignment Details: The study included a screening visit followed by visits every 4th week during dose escalation period and every 8th week until end-of-treatment (week 68). Follow-up period was 7 weeks after end-of-treatment (week 75).
Groups:
- Semaglutide 2.4 mg: Participants initiated at a once-weekly dose of 0.24 milligrams (mg) semaglutide subcutaneously (s.c.) as a adjunct to a reduced calorie diet and increased physical activity and followed a fixed-dose escalation regimen, with dose increase every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), until the target dose was reached after 16 weeks. Participants continued 2.4 mg semaglutide s.c. once- weekly from week 16 to week 68 as a adjunct to a reduced calorie diet and increased physical activity. Participants were followed up for 7 weeks after end of treatment till week 75.
- Placebo: Participants received semaglutide matching placebo subcutaneously once weekly as a adjunct to a reduced calorie diet and increased physical activity from week 0 to week 68. Participants were followed up for 7 weeks after end of treatment till week 75.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 271 | 136
Full Analysis Set (FAS) | 271 | 136
Safety Analysis Set (SAS) | 269 | 135
Completed | 246 | 122
Not Completed | 25 | 14
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Lost to Follow-up | 7 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Failing to Meet Randomization Requirements | 2 | 1
Not completed — Site Closure | 7 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants according to the intention-to-treat principle.
Groups:
- Semaglutide 2.4 mg: Participants initiated at a once-weekly dose of 0.24 mg semaglutide s.c. as a adjunct to a reduced calorie diet and increased physical activity and followed a fixed-dose escalation regimen, with dose increase every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), until the target dose was reached after 16 weeks. Participants continued 2.4 mg semaglutide s.c. once- weekly from week 16 to week 68 as a adjunct to a reduced calorie diet and increased physical activity. Participants were followed up for 7 weeks after end of treatment till week 75.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 271 | 136 | 407
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (10) | 56 (10) | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 104 | 332
  Male | 43 | 32 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 13 | 56
  Not Hispanic or Latino | 216 | 112 | 328
  Unknown or Not Reported | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 37 | 11 | 48
  Asian | 16 | 6 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 13 | 31
  White | 168 | 80 | 248
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 32 | 26 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Body Weight
Description: Percentage change in body weight from baseline (week 0) to end of treatment (week 68) is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: FAS included all randomized participants according to the intention-to-treat principle. Here, Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 253 | 120
Percentage change in body weight | -14.2 (8.6) | -2.5 (5.6)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; The responses at week 68 were analyzed using an analysis of covariance model with randomized treatment as factor and baseline body weight as covariate; Test type: Superiority; p < 0.0001, ANCOVA; Estimated Treatment Difference = -10.48, 95% CI 2-sided [-12.34 to -8.63]

2. Primary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score
Description: WOMAC is a disease-specific patient-reported outcome measure designed to assess changes in symptoms and lower extremity functioning associated with treatment in patients with osteoarthritis of the hip and/or knee. WOMAC is a 24 item questionnaire which assesses clinically important, participant-relevant symptoms in area of pain, stiffness, and physical function in participants with osteoarthritis (OA). It consists of 3 subscales: pain, stiffness and physical function. The WOMAC raw pain score is derived as the sum of the 5 item scores in the pain domain. It will be normalised and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the raw score for the pain domain (i.e. 50) and multiplying by 100. Higher scores indicate worse outcome. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 245 | 117
Score on a scale | -43.7 (25.3) | -26.2 (25.0)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; The responses at week 68 were analyzed using an analysis of covariance model with randomized treatment as factor and baseline WOMAC pain score as covariate; Test type: Superiority; p < 0.0001, ANCOVA; Estimated Treatment Difference = -14.14, 95% CI 2-sided [-19.98 to -8.30]

3. Secondary Outcome: Percentage of Participants Achieving Body Weight Reduction Greater Than or Equal to (≥) 5 Percent (%) (Yes/No)
Description: Percentage of participants who achieved ≥ 5% body weight reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥5% weight reduction whereas 'No' infers percentage of participants who have not achieved ≥5% weight reduction. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 253 | 120
Percentage of participants
  Yes | 87.0 | 29.2
  No | 13.0 | 70.8

4. Secondary Outcome: Percentage of Participants Achieving Body Weight Reduction ≥ 10% (Yes/No)
Description: Percentage of participants who achieved ≥10% body weight reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥10% weight reduction whereas 'No' infers percentage of participants who have not achieved ≥10% weight reduction. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 253 | 120
Percentage of participants
  Yes | 70.4 | 9.2
  No | 29.6 | 90.8

5. Secondary Outcome: Change in WOMAC Physical Function Score
Description: Change in WOMAC physical function score is presented. WOMAC is a 24 item questionnaire which assesses clinically important, participant-relevant symptoms in area of pain, stiffness, and physical function in participants with osteoarthritis (OA). It consists of 3 subscales: pain, stiffness and physical function. WOMAC physical function is 17-item questionnaire used to assess degree of difficulty experienced due to OA in knee. It is calculated as the sum of the 17 item scores in the physical function domain. It is normalized and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the raw score for the physical function domain (i.e. 170) and multiplying by 100. Higher scores indicate worse outcome. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: FAS included all randomized participants according to the intention-to-treat principle. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 117
Score on a scale | -43.4 (25.5) | -25.8 (25.1)

6. Secondary Outcome: Change in Short Form 36 (SF-36) Physical Functioning Score
Description: SF-36 is self-administered questionnaire that measures each of following 8 health domains: physical functioning, role limitations due to physical problems (role-physical), social functioning, bodily pain, mental health, role limitations due to emotional problems (role-emotional), vitality, and general health perception. There are also 2 component scores derived from the 8 subscale scores: physical component summary (including physical functioning, role-physical, bodily pain and general health) and mental component summary (including vitality, social functioning, role-emotional and mental health). Each SF-36 domain and component summary score ranges from 0 to 100, higher scores reflect better participant health status. A positive change score indicates an improvement since baseline. The outcome measure was evaluated based on data from in-trial period. In-trial period was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 241 | 115
Score on a scale | 12.7 (9.9) | 6.4 (9.8)

7. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to end of the treatment (visit 68) is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 253 | 120
Centimeter | -13.3 (9.3) | -5.9 (10.4)

8. Secondary Outcome: Change in WOMAC Stiffness Score
Description: WOMAC is a disease-specific patient-reported outcome measure designed to assess changes in symptoms and lower extremity functioning associated with treatment in patients with osteoarthritis of the hip and/or knee. WOMAC is a 24 item questionnaire which assesses clinically important, participant-relevant symptoms in area of pain, stiffness, and physical function in participants with OA. It consists of 3 subscales: pain, stiffness and physical function. The WOMAC raw stiffness score is derived as the sum of the 2 item scores in the stiffness domain. It will be normalized and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the raw score for the stiffness domain (i.e. 20) and multiplying by 100. Higher scores indicate worse outcome. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 117
Score on a scale | -45.4 (27.7) | -27.6 (29.3)

9. Secondary Outcome: Change in WOMAC Total Score
Description: WOMAC is a disease-specific patient-reported outcome measure designed to assess changes in symptoms and lower extremity functioning associated with treatment in patients with osteoarthritis of the hip and/or knee. WOMAC is a 24 item questionnaire which assesses clinically important, participant-relevant symptoms in area of pain, stiffness, and physical function in participants with OA. The WOMAC raw total score is derived as the sum of the 24 item scores respectively on pain, stiffness and physical function domain. It will be normalized and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the raw score for the total domain (i.e. 240) and multiplying by 100. Higher scores indicate worse outcome. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 245 | 117
Score on a scale | -43.8 (24.9) | -26.0 (24.9)

10. Secondary Outcome: Change in SF-36 Bodily Pain Score
Description: Change in SF-36 Bodily Pain Score from baseline (week 0) to end of treatment (week 68) is presented. SF-36 is self-administered questionnaire that measures each of following 8 health domains: physical functioning, role limitations due to physical problems (role-physical), social functioning, bodily pain, mental health, role limitations due to emotional problems (role-emotional), vitality, and general health perception. There are also 2 component scores derived from the 8 subscale scores: physical component summary and mental component summary. Each SF-36 domain and component summary score ranges from 0 to 100, higher scores reflect better participant health status. A positive change score indicates an improvement since baseline. The outcome measure was evaluated based on data from in-trial period. In-trial period was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 241 | 115
Score on a scale | 12.8 (9.4) | 7.7 (10.0)

11. Secondary Outcome: Change in SF-36 Physical Component Summary
Description: Change in SF-36 physical component summary is presented. It is self-administered questionnaire that measures each of following 8 health domains: physical functioning, role limitations due to physical problems (role-physical), social functioning, bodily pain, mental health, role limitations due to emotional problems (role-emotional), vitality, and general health perception. There are also 2 component scores derived from the 8 subscale scores: physical component summary and mental component summary. Physical component summary contains physical functioning, role-physical, bodily pain and general health. Each SF-36 domain and component summary score ranges from 0 to 100, higher scores reflect better participant health status. A positive change score indicates an improvement since baseline. The outcome measure was evaluated based on data from in-trial period. In-trial period was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 241 | 115
Score on a scale | 13.2 (9.1) | 6.9 (9.3)

12. Secondary Outcome: Change in SF-36 Mental Component Summary
Description: Change in SF-36 mental component summary is presented. SF-36 is self-administered questionnaire that measures each of following 8 health domains: physical functioning, role limitations due to physical problems (role-physical), social functioning, bodily pain, mental health, role limitations due to emotional problems (role-emotional), vitality, and general health perception. There are also 2 component scores derived from the 8 subscale scores: mental component summary and physical component summary. Mental component summary contain vitality, social functioning, role-emotional and mental health. Each SF-36 domain and component summary score ranges from 0 to 100, higher scores reflect better participant health status. A positive change score indicates an improvement since baseline. The outcome measure was evaluated based on data from in-trial period. In-trial period was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 241 | 115
Score on a scale | 1.9 (11.3) | 1.1 (11.6)

13. Secondary Outcome: Percentage of Participants Using Allowed Rescue Analgesics During Wash Out (Yes/No)
Description: Percentage of participants using allowed rescue analgesics during wash out at end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have used allowed rescue analgesics during wash out whereas 'No' infers percentage of participants who have not used allowed rescue analgesics during wash out. Use of allowed rescue analgesics is evaluated based on use of acetaminophen reported in the pain medication diary from one up to 3 days prior to WOMAC assessment. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: At end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 117
Percentage of participants
  Yes | 4.9 | 5.1
  No | 95.1 | 94.9

14. Secondary Outcome: Amount of Allowed Rescue Analgesics Used During Wash Out
Description: Amount of allowed rescue analgesics used during wash out at end of treatment (week 68) is presented. Allowed rescue analgesic during washout is defined as acetaminophen taken 24-72 hour before the visit. The outcome measure is approximated by a total dose of acetaminophen reported in the pain medication diary from one and up to 3 days prior to WOMAC assessment. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: At end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 117
Milligram | 224.2 (1756.4) | 170.1 (1100.3)

15. Secondary Outcome: Percentage of Participants With Use of Pain Medication
Description: Percentage of participants with use of pain medication from baseline (week 0) to end of treatment (week 68) is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: FAS included all randomized participants according to the intention-to-treat principle.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 271 | 136
Percentage of participants
  Opioids | 8.5 | 9.6
  NSAID | 55.7 | 59.6
  Acetaminophen | 57.2 | 58.1

16. Secondary Outcome: Change in Pain Intensity (Numerical Rating Scale [NRS])
Description: Pain intensity was assessed on an 11-point NRS over the past 24 hours (before each specified visit), where a score of 0 indicated "no pain" and a score of 10 indicated "worst possible pain", where higher the score, greater the pain intensity. Response at visit was derived from the pain diary data as an average score over 4 days interval leading up to visit-related washout period for pain medication. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), end of treatment (week 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 199 | 82
Score on a scale | -2.9 (2.7) | -1.4 (2.4)

17. Secondary Outcome: Percentage of Participants Achieving Body Weight Reduction ≥ 15% (Yes/No)
Description: Percentage of participants who achieved ≥15% body weight reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥15% weight reduction whereas 'No' infers percentage of participants who have not achieved ≥15% weight reduction. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 253 | 120
Percentage of participants
  Yes | 47.8 | 2.5
  No | 52.2 | 97.5

18. Secondary Outcome: Percentage of Participants Achieving Body Weight Reduction ≥ 20% (Yes/No)
Description: Percentage of participants who achieved ≥20% body weight reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥20% weight reduction whereas 'No' infers percentage of participants who have not achieved ≥20% weight reduction. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 253 | 120
Percentage of participants
  Yes | 23.3 | 0
  No | 76.7 | 100

19. Secondary Outcome: Percentage of Participants Achieving WOMAC Pain Reduction ≥ 30% (Yes/No)
Description: Percentage of participants who achieved ≥30% WOMAC pain reduction (yes/no) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥30% WOMAC pain reduction whereas 'No' infers percentage of participants who have not achieved ≥30% WOMAC pain reduction. WOMAC raw pain score is derived as sum of 5 item scores in pain domain. It will be normalized and expressed on 0-100 scale. This is done by dividing raw score by highest possible value of raw score for pain domain (i.e. 50) and multiplying by 100. Higher scores indicate worse outcome. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 245 | 117
Percentage of participants
  Yes | 78.8 | 56.4
  No | 21.2 | 43.6

20. Secondary Outcome: Percentage of Participants Achieving WOMAC Pain Reduction ≥ 50% (Yes/No)
Description: Percentage of participants who achieved ≥50% WOMAC pain reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥50% WOMAC pain reduction whereas 'No' infers percentage of participants who have not achieved ≥50% WOMAC pain reduction. WOMAC raw pain score is derived as sum of 5 item scores in pain domain. It will be normalized and expressed on 0-100 scale. This is done by dividing raw score by highest possible value of raw score for pain domain (i.e. 50) and multiplying by 100. Higher scores indicate worse outcome. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 245 | 117
Percentage of participants
  Yes | 66.9 | 34.2
  No | 33.1 | 65.8

21. Secondary Outcome: Percentage of Participants Achieving Threshold for Clinically Meaningful Within-participant Change in WOMAC Pain Score (Yes/No)
Description: Percentage of participants who achieved threshold for clinically meaningful within-participant change in WOMAC pain score from baseline (week 0) to end of treatment (week 68) is presented. The threshold refers to the decrease of at least 37.3 in the WOMAC pain score and it is derived based on 1-category improvement on patient global impression of status (PGI-S) scale. In reported data, 'Yes' infers percentage of participants who have achieved threshold whereas 'No' infers percentage of participants who have not achieved threshold. WOMAC raw pain score is derived as sum of 5 item scores in pain domain. It will be normalized and expressed on 0-100 scale. This is done by dividing raw score by highest possible value of raw score for pain domain (i.e. 50) and multiplying by 100. Higher scores=worse outcome. Outcome measure was evaluated based on data from in-trial period and it was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 245 | 117
Percentage of participants
  Yes | 61.2 | 33.3
  No | 38.8 | 66.7

22. Secondary Outcome: Percentage of Participants Achieving Threshold for Clinically Meaningful Within-participant Change in WOMAC Physical Function Score (Yes/No)
Description: Percentage of participants who achieved threshold for clinically meaningful within-participant change in WOMAC physical function score from baseline (week 0) to end of treatment (week 68) is presented. The threshold refers to the decrease of at least 41.2 in the WOMAC physical function score and it is derived based on 1-category improvement on PGI-S scale. In reported data, 'Yes' infers percentage of participants who have achieved threshold whereas 'No' infers percentage of participants who have not achieved threshold. WOMAC raw pain score is derived as sum of 5 item scores in pain domain. It will be normalized and expressed on 0-100 scale. This is done by dividing raw score by highest possible value of raw score for pain domain (i.e. 50) and multiplying by 100. Higher scores indicate worse outcome. Outcome measure was evaluated based on data from in-trial period and it was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 117
Percentage of participants
  Yes | 54.1 | 29.1
  No | 45.9 | 70.9

23. Secondary Outcome: Percentage of Participants Achieving Threshold for Clinically Meaningful Within-participant Change in SF-36 Physical Functioning Score (Yes/No)
Description: Percentage of participants who achieved threshold for clinically meaningful within-participant change in SF-36 physical function score is presented. Threshold refers to increase of at least 11.4 in SF-36 physical functioning score & it is derived based on 1-category improvement on PGI-S scale. 'Yes' infers percentage of participants who achieved threshold; 'No' infers percentage of participants who have not achieved threshold. SF-36: self-administered questionnaire that measures each of following 8 health domains: physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, & general health perception. Each SF-36 domain and component summary score ranges from 0-100, higher scores mean better participant health status. Outcome measure was evaluated based on data from in-trial period: uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 241 | 115
Percentage of participants
  Yes | 60.6 | 28.7
  No | 39.4 | 71.3

24. Secondary Outcome: Percentage of Participants Achieving Pain Intensity (Numerical Rating Scale [NRS]) Reduction ≥ 30% (Yes/No)
Description: Percentage of participants who achieved ≥30% pain intensity reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥30% pain intensity reduction whereas 'No' infers percentage of participants who have not achieved ≥30% pain intensity reduction. Response at visit was derived from the pain diary data as an average score over 4 days interval leading up to visit-related washout period for pain medication. Pain intensity was assessed on an 11-point NRS over the past 24 hours (before each specified visit), where a score of 0 indicated "no pain" and a score of 10 indicated "worst possible pain", where higher the score, greater the pain intensity. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 199 | 82
Percentage of participants
  Yes | 64.8 | 39.0
  No | 35.2 | 61.0

25. Secondary Outcome: Percentage of Participants Achieving Pain Intensity (Numerical Rating Scale [NRS]) Reduction ≥ 50% (Yes/No)
Description: Percentage of participants who achieved ≥50% pain intensity reduction (yes/no) from baseline (week 0) to end of treatment (week 68) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved ≥50% pain intensity reduction whereas 'No' infers percentage of participants who have not achieved ≥50% pain intensity reduction. Response at visit was derived from the pain diary data as an average score over 4 days interval leading up to visit-related washout period for pain medication. Pain intensity was assessed on an 11-point NRS over the past 24 hours (before each specified visit), where a score of 0 indicated "no pain" and a score of 10 indicated "worst possible pain", where higher the score, greater the pain intensity. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 68)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 199 | 82
Percentage of participants
  Yes | 49.7 | 28.0
  No | 50.3 | 72.0

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to end of trial (week 75)
Description: All presented adverse events are treatment-emergent adverse events (TEAEs). A TEAEs was defined as an event that had onset during the on-treatment period (date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least two consecutive missed doses). SAS included all randomized participants exposed to at least one dose of randomized treatment.
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/269 | 0/135
Serious Adverse Events (participants affected / at risk) | 27/269 | 11/135
Other Adverse Events (participants affected / at risk) | 128/269 | 51/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=269) | Placebo (N=135)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric pH decreased (Investigations) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmodium malariae infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Sleeve gastrectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=269) | Placebo (N=135)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 13 (13)
COVID-19 (Infections and infestations) | 50 (54) | 30 (31)
Constipation (Gastrointestinal disorders) | 32 (35) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 21 (32) | 7 (8)
Headache (Nervous system disorders) | 16 (18) | 5 (5)
Nausea (Gastrointestinal disorders) | 59 (109) | 12 (16)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 7 (8)
Vomiting (Gastrointestinal disorders) | 21 (30) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT05064735/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT05064735/SAP_002.pdf